CLINICAL TRIAL: NCT04337242
Title: Blended Care Psychodynamic Therapy or Cognitive Behavioral Therapy Versus Face-to-Face Psychotherapy for Depression: A Pragmatic Multicenter Randomized Controlled Non-inferiority Trial
Brief Title: Blended Care Versus Face-to-Face Therapy for Depression
Acronym: BLENDED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Belgium Health Care Knowledge Centre (Other Government); Erasmus University Rotterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S59765
Record Dates: First submitted 2020-02-11; First posted 2020-04-07 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder
Keywords: depression; psychotherapy; blended; cognitive behavioral; psychodynamic
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blended Dynamic Interpersonal Therapy (B-DIT) (Experimental): B-DIT is based on the same treatment principles as face-to-face Dynamic Interpersonal Therapy (DIT) and has the same structure of treatment consisting of three phases: (a) an exploration and engagement phase, (b) a middle or working through phase, and (c) an ending phase. B-DIT consists of 8 online modules that are alternated with up to 8 fortnightly face-to-face sessions.
  Interventions: Behavioral: B-DIT
- Blended Cognitive Behavioral Therapy (B-CBT) (Experimental): B-CBT is based on the same treatment principles as face-to-face Cognitive Behavioral Therapy (CBT). These include (a) psycho-education about depression, (b) cognitive restructuring (i.e., identifying and challenging maladaptive thoughts and beliefs, fostering problem solving capacities), (c) mindfulness and acceptance based approaches, and (d) relapse prevention. B-CBT in this trial consists of 8 online modules that are alternated with up to 8 fortnightly face-to-face sessions.
  Interventions: Behavioral: B-CBT
- Dynamic Interpersonal Therapy (DIT) (Active Comparator): DIT is a short-term, integrative psychodynamic, 16 weekly sessions individual therapy for depression. DIT formulates the presenting symptoms of depression as responses to interpersonal difficulties or perceived threats to attachments (loss/separation) and hence also as threats to the self.
  Interventions: Behavioral: DIT
- Cognitive Behavioral Therapy (CBT) (Active Comparator): CBT is a brief talking therapy that consists of a maximum of 16 sessions, offered over 4 to 6 months. CBT is based on the assumption that depression is directly related to patterns of thinking. Specifically, dysfunctional and often automatic patterns of thinking are assumed to be related to the onset and maintenance of depression.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: B-DIT — Blended Dynamic Interpersonal Therapy
  Arms: Blended Dynamic Interpersonal Therapy (B-DIT)
Behavioral: B-CBT — Blended Cognitive Behavioral Therapy
  Arms: Blended Cognitive Behavioral Therapy (B-CBT)
Behavioral: DIT — Dynamic Interpersonal Therapy
  Arms: Dynamic Interpersonal Therapy (DIT)
Behavioral: Cognitive Behavioral Therapy — CBT
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
Depression is a severe mental disorder that affects 5-7% of Belgians each year. Unfortunately, many individuals with depression do not seek professional help, and if they do seek professional help, waiting lists for psychotherapy are typically very long.

To help resolve this problem, this study aims to investigate whether blended therapies, i.e. therapies that consist of a mixture of face-to-face sessions and online sessions, are (cost-)effective as a treatment for depression, and whether they are as (cost-)effective as traditional treatments which consist of face-to-face sessions alone. Should this be the case, then blended therapy can be implemented on a large scale in mental health care, as it could provide a more cost-effective means of helping individuals with depression.

This study also aims to investigate whether certain patient features, such as the severity of depression and personality traits, may influence the efficacy of (blended) psychotherapy for depression.

Finally, we will also investigate patients' attitudes towards and experience of blended therapy.

DETAILED DESCRIPTION:
Depression is a highly prevalent disorder with a lifetime prevalence of 15-25%, and is associated with high psychosocial and economic costs (e.g, suicide, absenteeism, long-term disability). Epidemiological research shows that depression is underrecognized and underdiagnosed in Belgium, resulting in very high unmet needs, with more than 50% of patients not seeking professional help in the first year after onset and often taking patients up to 10 years and more to effectively seek professional help (Bruffaerts et al., 2007, 2008). The current lack of capacity of mental health services in Belgium is a major obstacle in attempts to increase access to effective psychotherapy for depression. Centers for Mental Health Care ('Centra Geestelijke Gezondheidszorg', CGGs) in particular are faced with a growing number of patients (+3% per year). Despite their efforts (e.g., by offering more group-based psychotherapy and interventions), CGGs in Belgium are faced with increasingly longer waiting lists. There is therefore an urgent need for (cost-)effective, time-saving interventions in the mental health care system in Belgium.

Both pharmacotherapy and psychotherapy alone or in combination have been shown to be effective in the treatment of depression, and meta-analyses have shown no substantial differences in the efficacy of two of the empirically most validated types of brief face-to-face (FTF) psychotherapy in major depression, i.e., Cognitive Behavioral Therapy (CBT) and Psychodynamic Therapy (PDT) (Cuijpers et al., 2013; Cuijpers, Van Straten, Van Oppen, & Andersson, 2008; Driessen et al., 2015; Luyten & Blatt, 2012; Munder et al., 2018). Moreover, meta-analyses and qualitative reviews converge to suggest that internet-based interventions, particularly offered as blended care (combining face-to-face sessions with internet-based modules), may be equally effective as FTF psychotherapy and pharmacotherapy in major depression both at treatment termination and at follow-up in the medium to long-term, suggesting non-inferiority (Andersson, Cuijpers, Carlbring, Riper, & Hedman, 2014). Extant research in this domain also suggests that both CBT and PDT delivered through the internet may be effective in depression. Moreover, the available evidence suggests that internet-based psychotherapy if combined with therapist support may be more cost-effective as it typically reduces the number of face-to-face contacts, without compromising the effectiveness of psychotherapy (Andersson, Titov, Dear, Rozental, & Carlbring, 2019). Hence, the implementation of blended care may lead to increased availability of psychotherapy for depression and a more effective use of resources in mental health care, at least for a subsample of depressed patients.

The primary objective of this study is therefore to investigate the non-inferiority (defined as a small-sized difference in effect size (Cohen's d= .20) of blended PDT and CBT for depression compared to FTF PDT and CBT in adults diagnosed with major depressive disorder (n=504) in the context of a pragmatic, multicenter randomized controlled trial. Patients will be randomized to one of four conditions (i.e., blended PDT, blended CBT, FTF PDT, or FTF CBT). The primary outcome is changes in the severity of depression as measured by the Beck Depression Inventory (BDI-II; Beck, Steer, & Brown, 1996) at 6 months follow-up (approximately 12 months after the start of treatment).

In addition, this study will investigate the comparative efficacy of blended care versus FTF psychotherapy on the following secondary outcomes: severity of depression as measured with the BDI-II at treatment termination, and at 6-month, and one- and two-year follow-up; recovery from depression as assessed with the Structured Clinical Interview for DSM 5 disorders - Clinical Trials Version (SCID-5-CT; American Psychiatric Association) and the Patient Health Questionnaire-9 (PHQ-9) at treatment termination, and at 6-month, and one- and two-year follow-up; and quality of life as measured with the EuroQol-5D-5L (EQ-5D-5L; Herdman et al., 2011) at treatment termination, and at 6-month, and one- and two-year follow-up.

Furthermore, this study will also examine possible predictors of treatment response in blended care versus FTF therapy, such as severity of depression (BDI-II, PHQ-9), psychiatric co-morbidity (SCID-5-CT), and patients' experience of both types of treatment as assessed with the Credibility and Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000). In addition, the feasibility of implementing blended care in mental health care centers in Flanders, Belgium, will be investigated. To this end, we will record recruitment rate, retention in treatment, treatment adherence, and adherence to the research protocol. Acceptability will be indicated by the number of sessions attended, including the number of individuals who refuse treatment, and feasibility by the number of patients failing to comply with the full clinical and research protocol. Patients will also complete very brief measures of credibility of the treatments and satisfaction with the treatments. Treatment integrity of therapists will be assessed on the basis of independent ratings of audio or video recorded psychotherapy sessions, applying a treatment integrity instrument developed in the UK specifically for the treatments used in this study (Lemma, Target, & Fonagy, 2011).

Finally, provided blended care is non-inferior to FTF therapy, the cost-effectiveness of blended care versus FTF psychotherapy will be investigated from a societal perspective, i.e., taking all relevant costs and effects into account (intervention costs, direct and indirect medical costs, as well as productivity losses and costs made elsewhere in the health care system). To this end, patients will complete the Trimbos and Institute for Medical Technology Assessment (iMTA) Questionnaire on Costs Associated with Psychiatric Illness (TIC-P; Bouwmans et al., 2013). Moreover, health care use data for all patients will be provided by the Rijksinstituut voor Ziekte- en Invaliditeitsverzekering (RIZIV).

References

Andersson, G., Cuijpers, P., Carlbring, P., Riper, H., & Hedman, E. (2014). Guided Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: a systematic review and meta-analysis. World Psychiatry, 13(3), 288-295. doi:10.1002/wps.20151

Andersson, G., Titov, N., Dear, B. F., Rozental, A., & Carlbring, P. (2019). Internet-delivered psychological treatments: from innovation to implementation. World Psychiatry, 18(1), 20-28. doi:10.1002/wps.20610

Beck, A., Steer, R., & Brown, G. (1996). Manual for Beck Depression Inventory - II (BDI-II). San Antonia, TX: Psychological Corporation.

Bouwmans, C., De Jong, K., Timman, R., Zijlstra-Vlasveld, M., Van der Feltz-Cornelis, C., Tan, S. S., & Hakkaart-van Roijen, L. (2013). Feasibility, reliability and validity of a questionnaire on healthcare consumption and productivity loss in patients with a psychiatric disorder (TiC-P). BMC Health Services Research, 13, 217-217. doi:10.1186/1472-6963-13-217

Bruffaerts, R., Bonnewyn, A., & Demyttenaere, K. (2007). Delays in seeking treatment for mental disorders in the Belgian general population. Social Psychiatry and Psychiatric Epidemiology, 42(11), 937-944. doi:10.1007/s00127-007-0239-3

Bruffaerts, R., Bonnewyn, A., & Demyttenaere, K. (2008). Het voorkomen van depressie in België. Stand van zaken en reflecties voor de toekomst. Tijdschrift voor Psychiatrie, 50(10), 655-665.

Cuijpers, P., Berking, M., Andersson, G., Quigley, L., Kleiboer, A., & Dobson, K. S. (2013). A meta-analysis of cognitive-behavioural therapy for adult depression, alone and in comparison with other treatments. Canadian Journal of Psychiatry, 58(7), 376-385.

Cuijpers, P., Van Straten, A., Van Oppen, P., & Andersson, G. (2008). Are psychological and pharmacologic interventions equally effective in the treatment of adult depressive disorders? A meta-analysis of comparative studies. Journal of Clinical Psychiatry, 69(11), 1675-1685.

Devilly, G. J., & Borkovec, T. D. (2000). Psychometric properties of the credibility/expectancy questionnaire. Journal of Behavior Therapy and Experimental Psychiatry, 31(2), 73-86.

Driessen, E., Hegelmaier, L. M., Abbass, A. A., Barber, J. P., Dekker, J. J., Van, H. L., . . . Cuijpers, P. (2015). The efficacy of short-term psychodynamic psychotherapy for depression: A meta-analysis update. Clinical Psychology Review, 42, 1-15. doi:10.1016/j.cpr.2015.07.004

Herdman, M., Gudex, C., Lloyd, A., Janssen, M., Kind, P., Parkin, D., . . . Badia, X. (2011). Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Quality of Life Research, 20(10), 1727-1736. doi:10.1007/s11136-011-9903-x

Lemma, A., Target, M., & Fonagy, P. (2011). Brief dynamic interpersonal therapy. A clinician's guide. Oxford: Oxford University Press.

Luyten, P., & Blatt, S. J. (2012). Psychodynamic treatment of depression. Psychiatric Clinics of North America, 35(1), 111-129.

Munder, T., Fluckiger, C., Leichsenring, F., Abbass, A. A., Hilsenroth, M. J., Luyten, P., . . . Wampold, B. E. (2018). Is psychotherapy effective? A re-analysis of treatments for depression. Epidemiol Psychiatr Sci, 1-7. doi:10.1017/s2045796018000355 1-7. doi:10.1017/s2045796018000355

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Current diagnosis of major depressive disorder with or without dysthymic disorder according to DSM 5 criteria.
* PHQ score ≥ 10.

Note: Use of pharmacotherapy for depression and other psychiatric disorders during the intervention is allowed (with the exception of antipsychotic medication for psychotic disorder), as this reflects routine clinical care. Of note, in routine clinical care, it is not uncommon that antipsychotic medication is prescribed for symptoms in the depressive-anxious cluster rather than for primary psychotic symptoms.

Exclusion Criteria:

* Current psychotic symptoms or bipolar disorder.
* Current use of antipsychotic medication specifically for the treatment of primary psychotic disorder.
* Severe Personality Disorder (e.g., borderline personality disorder).
* Historic or current self-injury/parasuicide of such extent and/or severity that may substantially interfere with the ability to engage in brief psychotherapy.
* Current excessive use of drugs/alcohol.
* Not fluent in Dutch.
* Clinical contra-indication to brief psychotherapy (e.g., attachment history - multiple separations, serious ongoing trauma in childhood, multiple caregivers - suggesting the need for longer-term psychotherapy).
* Evidence of pervasive use of help.
* Highly unstable or insecure life arrangements.
* No access to computer/internet or computer illiteracy.
* Participation in another depression clinical trial within the last year where the participant has received CBT or PDT.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in depressive symptoms assessed by the Beck Depression Inventory (BDI-II) at 6-month follow-up (12 months after the start of treatment) | From baseline to 6 months follow-up (12 months after the start of treatment)
  Severity of depression as measured by the BDI-II (range 0-63, with higher scores reflecting worse outcome)

SECONDARY OUTCOMES:
Partial and full recovery | From baseline to treatment termination (6 months after the start of treatment), and 6-month, and one- and two-year follow-up
  Full recovery as assessed with the Structured Clinical Interview for DSM 5 disorders - Clinical Trials Version (SCID-5-CT) is defined as at least two consecutive months in which no MDD symptoms were present, partial recovery as assessed with the Structured Clinical Interview for DSM 5 disorders - Clinical Trials Version (SCID-5-CT) as maximum 1-4 symptoms of MDD present in the last two months.
  Full recovery as assessed with the Patient Health Questionnaire-9 (PHQ-9) is defined as scoring below 4, partial recovery as scoring between 5-9.
Quality of Life | From baseline to treatment termination(6 months after the start of treatment), and 6-month, and one- and two-year follow-up
  Quality of Life as measured with the EuroQol-5D-5L. The EQ-5D-5L measures quality of life in five dimensions of health (mobility, self-help, habitual activities, pain, anxiety/depression), each with five levels reflecting "no problems", "slight problems", "moderate problems", "severe problems", and "extreme problems". The EQ Visual Analogue Scale in turn records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labeled 'the best health you can imagine' and 'the worst health you can imagine'.
Treatment Expectancy | Baseline, and (with a modified version) at treatment termination (6 months after the start of treatment) and 6-month follow-up
  Patients' expectancy of treatment will be measured with the Credibility and Expectancy Questionnaire (CEQ)
Satisfaction with treatment | Baseline, treatment termination (6 months after the start of treatment), and at 6-month, and one- and two-year follow-up
  Satisfaction of patients with treatment as assessed by the Client Satisfaction Questionnaire-8 (CSQ-8)
Cost-effectiveness | Baseline, treatment termination (6 months after the start of treatment), and at 6-month, and one- and two-year follow-up
  Cost-effectiveness will be analyzed using the Trimbos and Institute for Medical Technology Assessment (iMTA) Questionnaire on Costs Associated with Psychiatric Illness (TIC-P) and health care data provided by the Belgian Rijksdienst Voor Ziekte- en InvaliditeitsVerzekering (RIZIV) using a Markov model to project future costs and effects using different time horizons. We will also calculate detailed cost-effectiveness planes of the incremental costs in relation to gained QALYs at different willingness-to-pay thresholds.

OTHER OUTCOMES:
Predictors of treatment response and mechanisms of change | Baseline
  Patient features that have often been linked to negative treatment outcome, such as self-criticism and dependency measured with the Depressive Experiences Questionnaire (DEQ), severity of depression (BDI-II, PHQ-9), psychiatric co-morbidity as measured with the SCID interview, and patients' experience of both types of treatment as assessed with the Credibility and Expectancy Questionnaire (CEQ) will be examined
Feasibility and acceptability of blended psychotherapy | Baseline, treatment termination (6 months after the start of treatment), and at 6-month, and one- and two-year follow-up
  Recruitment rate, retention in treatment, treatment adherence, and adherence to the research protocol will be assessed throughout the trial. Acceptability will be indicated by the number of sessions attended, including the number of individuals who refuse treatment and feasibility by the number of patients failing to comply with the full clinical and research protocol. Treatment integrity of therapists will be assessed on the basis of independent ratings of audio or video recorded psychotherapy sessions. In addition, to measure patient attitudes towards the treatment programs, we will administer the Credibility and Expectancy Questionnaire (CEQ) at baseline and an adapted version of this measure at post-treatment and 6-month follow-up. Satisfaction with treatment will be measured with the Client Satisfaction Questionnaire-8 (CSQ-8).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Luyten, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (6):
- Belgium (6):
  - CGG Andante, Berchem
  - CGG Vagga, Berchem
  - CGG Mandel & Leie, Kortrijk
  - CGG VBO, Leuven
  - CGG De Pont, Mechelen
  - CGG Kempen, Turnhout

IPD SHARING:
Plan to Share IPD: Yes
The study results will be owned by the Sponsor. The sponsor will have access to the study data. At the end of the study, KCE will receive from the Sponsor specific study data. This will only be coded data made available to KCE.
  The study data shall not be provided to a third party without the prior written approval of KCE, which approval KCE shall not unreasonably withhold or delay and which KCE may subject to specific conditions in order to ensure that the provision of said study data does not have a negative impact on the further performance of the study, the rights granted to KCE under the research agreement and/or the benefit of the Study for the patients and/or the public payers. After the publication of results focusing on primary and secondary outcomes/endpoints, anonymous data will be made available to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the publication of results focusing on primary and secondary outcomes/endpoints, anonymous data will be made available.
Access Criteria: Only researchers who provide a methodologically sound research proposal can ask for access to the data.